CLINICAL TRIAL: NCT00372658
Title: Intracervical Block and Pain Perception During the Performance of a Hysterosalpingogram: A Randomized Controlled Trial
Brief Title: Intracervical Block Versus Placebo to Assess Pain Control During Hysterosalpingogram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20010125H
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2006-09-07 (Estimated); Status verified 2005-12

CONDITIONS: Infertility
Keywords: hysterosalpingogram; intracervical local anesthesia; pain perception; visual analogue scale
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Drug: 1% Lidocaine intracervical injection

SUMMARY:
The purpose of this study is to compare the efficacy of 1% lidocaine intracervical block to placebo for pain control during the performance of a hysterosalpingogram (HSG). We hypothesized that an intracervical block would decrease pain during a hysterosalpingogram.

DETAILED DESCRIPTION:
The hysterosalpingogram (HSG) is an integral part of the evaluation for anatomic etiologies of female infertility. The majority of women regard a hysterosalpingogram as acutely painful since it involves placement of a cervical tenaculum, traction on the cervix, and instillation of dye through a cervical cannula. Different techniques have been employed to attempt to make the procedure less painful, including use of balloon catheters rather than cannulas; however, this has not been shown to be uniformly effective. Previous studies have shown a reduction in overall pain during HSG after pre-medication with oral non-steroidal anti-inflammatory drugs. Benzocaine gel (20%) applied to the cervix has also been shown to reduce pain. Conversely, a study of pre-medication with paracetamol (acetaminophen) showed no statistical improvement in pain perception. Additionally, transcervical intrauterine instillation of lidocaine has been shown in randomized studies to not improve pain scores and may actually increase pain after the procedure is complete A MEDLINE literature search of papers written in English from January 1966 to August 2005, using the keywords "hysterosalpingogram," "analgesia", "paracervical," and "intracervical" did not reveal any prior studies on the use of an intracervical block prior to hysterosalpingography. A paracervical block has been shown to decrease pain with therapeutic abortions, endometrial biopsy, and office hysteroscopy (7, 8). We hypothesized that an intracervical block would also decrease pain during a hysterosalpingogram. A three armed, randomized controlled trial comparing pain control after a 1% lidocaine intracervical block, saline injection or no injection in patients undergoing hysterosalpingogram was performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients without a known cause for their infertility who were undergoing a hysterosalpingogram were eligible for enrollment.
* All subjects were 18 to 40 years of age and married.

Exclusion Criteria:

* Included a history of any allergies to local anesthetics, radio-opaque dye or to anti-inflammatory medications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2002-07; Study Completion 2004-10

PRIMARY OUTCOMES:
Visual analogue and qualitative scales to assess study participants pain at 6 different time points during the hysterosalpingogram.

SECONDARY OUTCOMES:
Anatomical result of the hysterosalpingogram were also collected for a sub-group analysis to evaluate if particular pathology had an effect on pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Randal D Robinson, MD, Principal Investigator — Wilford Hall Medical Center and Brooke Army Medical Center
Locations (1):
- Wiford Hall Medical Center, Lackland Air Force Base, Texas, United States

REFERENCES:
- [Derived] Robinson RD, Casablanca Y, Pagano KE, Arthur NA, Bates GW, Propst AM. Intracervical block and pain perception during the performance of a hysterosalpingogram: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):89-93. doi: 10.1097/01.AOG.0000247645.52211.41. PMID 17197592